CLINICAL TRIAL: NCT06871020
Title: Evaluation of Periodontal Health and Patient Satisfaction of CAD/CAM Fiber-Reinforced Composite Versus Porcelain Fused to Metal Extracoronal Attachment in Mandibular Distal Extension Removable Partial Dentures: A Randomized Clinical Trial
Brief Title: Periodontal Health and Patient Satisfaction of CAD/CAM Fiber-Reinforced vs. PFM Attachments in Distal Extension RPDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnia M. Refai, Lecturer of Oral and Maxillofacial Prosthodontics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-RecIR122439
Record Dates: First submitted 2025-02-22; First posted 2025-03-11 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-03

CONDITIONS: Mandibular Distal-extension Prostheses
Keywords: CAD/CAM; Fiber Reinforced Composite; Denture Precision Attachment; Denture, Partial, Removable

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OT Extracoronal attachment made from CAD-CAM fiber-reinforced composite resin. (Experimental): The patient will receive a removable partial denture retained by bilateral OT extracoronal attachments made from CAD/CAM fiber-reinforced composite resin. These attachments will be fabricated on the prepared first premolars and canines on each side.
  Interventions: Other: Mandibular removable partial denture retained on OT extracoronal attachment made from fiber-reinforced composite resin
- OT Extracoronal attachment made from porcelain-fused-to-metal (Active Comparator): The patient will receive a removable partial denture retained by bilateral T Extracoronal attachment made from porcelain-fused-to-metal . These attachments will be fabricated on the prepared first premolars and canines on each side.
  Interventions: Other: Mandibular removable partial denture retained on OT extracoronal attachment made from porcelain-fused to metal

INTERVENTIONS:
Other: Mandibular removable partial denture retained on OT extracoronal attachment made from fiber-reinforced composite resin — Bilateral OT extracoronal attachments will be milled from fiber-reinforced composite resin after obtaining impressions of the prepared abutments. This will be followed by an overall impression of fabricating a Co-Cr removable partial denture to be retained in the attachments.
  Arms: OT Extracoronal attachment made from CAD-CAM fiber-reinforced composite resin.
Other: Mandibular removable partial denture retained on OT extracoronal attachment made from porcelain-fused to metal — Bilateral OT attachments manufactured from porcelain fused to metal by conventional technique after obtaining impressions of the prepared abutments. This will be followed by an overall impression of fabricating a Co-Cr removable partial denture to be retained in the attachments.
  Arms: OT Extracoronal attachment made from porcelain-fused-to-metal

SUMMARY:
This randomized clinical trial aims to assess periodontal health and patient satisfaction in mandibular distal extension removable partial dentures using CAD/CAM fiber-reinforced composite versus porcelain-fused-to-metal extracoronal attachments. Twelve participants with bilateral mandibular Kennedy Class I, retaining only the first premolars as the last standing abutments, will be randomly assigned to two groups. Group I will receive OT extracoronal attachments made from CAD/CAM fiber-reinforced composite, while Group II will receive OT extracoronal attachments made from porcelain-fused-to-metal. All participants will then receive a metallic removable partial denture. The null hypothesis states that no significant differences will be observed in periodontal health and patient satisfaction between the two attachment types.

DETAILED DESCRIPTION:
Twelve participants with bilateral maxillary Kennedy Class I, with the first premolars as the last standing abutments, will be recruited based on strict inclusion criteria from the oral and maxillofacial prosthodontic outpatient clinic. The canines and first premolars will be prepared to receive OT extracoronal attachments made from either CAD/CAM fiber-reinforced composite (Group I) or porcelain-fused-to-metal (Group II), according to group allocation. All participants will then receive a metallic removable partial denture. Periodontal health will be assessed through bleeding index, probing depth, and gingival recession at denture insertion and after six months. Patient satisfaction will also be evaluated at the six-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Mandibular partially edentulous bilateral distal extension Kennedy Class I with first premolars as last abutments.
2. The opposing maxillary arch will be dentate.
3. Angle class I maxillomandibular skeletal relation.
4. The distal extension ridge will be well-formed and covered by healthy and firm mucosa.
5. As verified by periapical radiographs, Abutments have healthy periodontal ligaments and an appropriate crown/root ratio (CRR).
6. Crown/root ratio of the premolar abutment teeth is not less than 1:1. 5.
7. The vertical distance between the ridge tissue and the opposing teeth of the study cases is not less than 7 mm. 6.
8. The buccolingual dimension of the abutment teeth is not less than 6 mm.

Exclusion Criteria:

1. Patients with any systemic disease that could affect the rate of bone resorption, which was confirmed by obtaining a through medical history.
2. Patients with parafunctional habits (bruxism and clenching).
3. Patients with any septic foci or impacted teeth as proved by panoramic radiograph, as well as patients with tilted or rotated abutments or soft tissue undercuts in areas that will be involved in the RDP design.
4. Patients with any TMJ problems.
5. Patients with any neuromuscular diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Bleeding index | At denture insertion ( baseline 0) and six months (180 days) after delivery of mandibular removable partial denture retained on double OT Extracoronal attachments
  The bleeding Index will be evaluated at denture insertion and after six months (180 days: Assessed using Mombelli's Bleeding Index, which scores bleeding on probing (BOP) from 0 (no bleeding) to 3 (heavy bleeding).
Evaluation of Probing Pocket Depth (PPD) | At denture insertion ( baseline 0) and six months (180 days) after delivery of mandibular removable partial denture retained on double OT Extracoronal attachments
  Evaluation of Probing Pocket Depth (PPD)will be evaluated at denture insertion and after six months: Measured on buccal and lingual aspects of the four abutments following the American Academy of Periodontology protocol. Six readings per abutment will be averaged.
Evaluation of Gingival Recession | At denture insertion ( baseline 0) and six months (180 days) after delivery of mandibular removable partial denture retained on double OT Extracoronal attachments
  Evaluation of Gingival Recession: Measured from the cemento-enamel junction (CEJ) to the gingival margin.
Evaluation Gingival Index (GI) | At denture insertion ( baseline 0) and six months (180 days) after delivery of mandibular removable partial denture retained on double OT Extracoronal attachments
  Evaluation of Gingival index: Evaluated using Löe and Silness (1963), scoring gingival inflammation from 0 (healthy) to 3 (severe inflammation with spontaneous bleeding).

SECONDARY OUTCOMES:
Evaluation of Patient Satisfaction | After six months (180 days) after delivery of mandibular removable partial denture retained on double OT Extracoronal attachments
  Patient satisfaction will be evaluated using the McGill Denture Satisfaction Questionnaire and a visual analog scale (VAS). Satisfaction will be measured across multiple aspects, including ease of cleaning, speech ability, comfort, esthetics, stability, mastication of various foods, masticatory efficiency, oral condition, and overall satisfaction. Patients will rate each item on a 0-100 scale, where 0 represents complete dissatisfaction and 100 indicates total satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Omnia M. Refai, PHD, Principal Investigator — Ain Shams Univeristy; Noha Helmy Hassan Nawar, PHD, Study Director — Ain Shams Univeristy; Heba A. Salama, PHD, Principal Investigator — Misr International University; Abdel Rahman Maged, PHD, Principal Investigator — Misr International University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No